CLINICAL TRIAL: NCT01252446
Title: Children With ADHD Symptoms: Comorbid Conditions, Cognitive and Social Performance
Acronym: NF ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Helse Fonna (Other)
Responsible Party: Nezla Duric, MD, Child and Adolesc. Psych., University of Bergen, Child and Adolescent Clinic Helse Fonna
Other Study IDs: 219.04 REK; 219.04(REK)
Record Dates: First submitted 2010-11-19; First posted 2010-12-03 (Estimated); Last update posted 2010-12-03 (Estimated); Status verified 2009-01

CONDITIONS: Comorbid Conditions; Social-demographic Profiles
Keywords: ICD 10; Attention-Deficit-Hyperactivity-Disorder (ADHD); Comorbidity; Social-demographic profile
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ADHD: The sample of 187 children and adolescent in the age of 6 to 17 years referred to the Child and Adolescent Clinic, Haugesund, Norway during the period of one year and diagnosed in ICD 10 system as ADHD.

SUMMARY:
This article reviews social-demographic variables (SDV) including interpersonal and academic and social performance in families and comorbid conditions(CC) which are the most associated with Attention-Deficit/Hyperactivity Disorder (ADHD)in the sample that has been confirmed diagnosis of ADHD and sample with the same symptoms but not confirmed diagnosis of ADHD.

There are no reports of this kind in the Norwegian population with ADHD.

DETAILED DESCRIPTION:
ADHD is one of the largest diagnostic groups in psychiatric health care for children and adolescents in Norway. In the guidelines laid out by the central authorities, ADHD is to be prioritized. As can be seen by the attention this topic is given in the media, good diagnostics and treatment for this group are important for society as well as the individuals who suffer from this. Early diagnosis, proper organization and appropriate treatment have a positive effect on the self-esteem and development of the person diagnosed as well as probable socio-economic benefits for society.

ADHD population shows significant pattern in socio-demographic relations and comorbidity according to the population that is referred to community Mental Health Clinic due another types of psychiatric conditions.

In terms of comorbid states ODD and OCD are most associated with ADHD . The study indicates prevalence of ADHD children (74%) who met criteria for ADHD, Combined Type (ADHD-C, both inattention and hyperactivity-impulsivity symptoms) and the existence of generally low IQ measures with mean value of 85 points. In terms of comorbid states generally were found in almost whole ADHD group (93 %) compared to half of the non-ADHD group. Disruptive Behaviour Disorder, Anxiety /Stress related disorder and Encopresis /Enuresis shows significant difference between the groups. Other comorbid conditions show no significant differences. Social dysfunctions were found in four of five children.

ELIGIBILITY:
Inclusion Criteria:

* clinical symptoms related on diagnosis of ADHD
* age from 6-17 years

Exclusion Criteria:

* retardation
* somatic disorder

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: One hundred eihgty seven children and adolescent referred to a Child and Adolescent Mental Health Clinic in Haugesund, Rogaland, Norway with the sympthoms of innattentivity, hyperactivity and impulsivity. Ninety one of them has been diagnosed with ADHD by the ICD 10 Classification and Diagnostic system and ninety six has been diagnised with other diagnosis accordning to ICD 10 classification .
  All referred children has been evaluated in this study. The diagnosis was made by child psychiatrist and relevant team and was based on the standard somatic and mental examination, information from the parents and teachers and diagnostics interviews.(Clinicians manual for assessment and parent training from Russell A. Barkley and SDQ-nor questionnaire ).
Sampling Method: Non-Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Clinicians Manuals from Russell A. Barkley as Disruptive Behavior Disorders Rating Scale--Parent Form (Form 4), Disruptive Behavior Disorders Rating Scale--Teacher Form (Form 5) and Clinical Interview--Parent Report Form (Form 6) | 1 year
  The population was selected from a specialized outpatient clinic for Child and Adolescent Mental Health in Norway. ADHD referred children were classified in two groups: ADHD and non-ADHD. The data was obtained by examination of children and adolescent and by personal interviews and questionnaire with parents, teachers, children and adolescent with attention-deficit/hyperactivity disorder (ADHD).

SECONDARY OUTCOMES:
cognitive performance | 1 year
  Wechsler Intelligence Scale for Children-Revised (WISC-R)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Elgen, m.d.PhD, Study Chair — University in Bergen; Nezla Duric, M.D., Principal Investigator — University in Bergen
Locations (1):
- Child and Adolescent Psychiatry Clinic Helse Fonna Haugesund, Haugesund, Rogaland, Norway

REFERENCES:
- [Background] Jensen PS, Hinshaw SP, Kraemer HC, Lenora N, Newcorn JH, Abikoff HB, March JS, Arnold LE, Cantwell DP, Conners CK, Elliott GR, Greenhill LL, Hechtman L, Hoza B, Pelham WE, Severe JB, Swanson JM, Wells KC, Wigal T, Vitiello B. ADHD comorbidity findings from the MTA study: comparing comorbid subgroups. J Am Acad Child Adolesc Psychiatry. 2001 Feb;40(2):147-58. doi: 10.1097/00004583-200102000-00009. PMID 11211363
- [Background] Pliszka SR. Psychiatric comorbidities in children with attention deficit hyperactivity disorder: implications for management. Paediatr Drugs. 2003;5(11):741-50. doi: 10.2165/00148581-200305110-00003. PMID 14580223
- [Background] da Silva MA, Louza MR, Vallada HP. Attention deficit hyperactivity disorder (ADHD) in adults: social-demographic profile from a university hospital ADHD outpatient unit in Sao Paulo, Brazil. Arq Neuropsiquiatr. 2006 Sep;64(3A):563-7. doi: 10.1590/s0004-282x2006000400004. PMID 17119791
- [Derived] Duric NS, Assmus J, Gundersen D, Elgen IB. Neurofeedback for the treatment of children and adolescents with ADHD: a randomized and controlled clinical trial using parental reports. BMC Psychiatry. 2012 Aug 10;12:107. doi: 10.1186/1471-244X-12-107. PMID 22877086
- See also: MTA study — http://www.ncbi.nlm.nih.gov/pubmed/17667478